CLINICAL TRIAL: NCT06610110
Title: Influence of CYP1A2 on the Acute Effect of Caffeine Intake on Resistance Exercise
Brief Title: Caffeine, CYPA12 and Resistance Exercise
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alberto Pérez-López (Other)
Collaborators: University of Alcala (Other); iSanidad+Herbalife (Unknown)
Responsible Party: Sponsor-Investigator, Alberto Pérez-López, Principal Investigator, University of Alcala
Organization: University of Alcala (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CEIP/2024/2/037
Record Dates: First submitted 2024-09-09; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: CYP1A2 Polymorphism; Caffeine and Resistance Exercise
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Genotype AA - Male - Caffeine (Experimental)
  Interventions: Dietary Supplement: Caffeine
- Genotype AC or CC - Male - Caffeine (Experimental)
  Interventions: Dietary Supplement: Caffeine
- Genotype AA - Male - Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Genotype AC or CC - Male - Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Genotype AA - Female - Caffeine (Experimental)
  Interventions: Dietary Supplement: Caffeine
- Genotype AC or CC - Female - Caffeine (Experimental)
  Interventions: Dietary Supplement: Caffeine
- Genotype AA - Female - Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Genotype AC or CC - Female - Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Caffeine — Acute caffeine intake (3 mg/kg)
  Arms: Genotype AA - Female - Caffeine; Genotype AA - Male - Caffeine; Genotype AC or CC - Female - Caffeine; Genotype AC or CC - Male - Caffeine
Dietary Supplement: Placebo — Placebo (3 mg/kg maltodextrin)
  Arms: Genotype AA - Female - Placebo; Genotype AA - Male - Placebo; Genotype AC or CC - Female - Placebo; Genotype AC or CC - Male - Placebo

SUMMARY:
Introduction: Several studies have evaluated and confirmed the ergogenic effect of acute caffeine intake on sports performance, specifically on strength and power performance. However, it remains to be elucidated how CYP1A2 polymorphism influences the acute effects of caffeine on this type of exercise.

Objectives: The present study aims to analyze the effects of acute caffeine intake on muscular strength, power, and endurance performance according to CYP1A2 polymorphism in men and women.

ELIGIBILITY:
Inclusion Criteria:

* Age between ≥ 18 and ≤ 35 years.
* Body mass index (BMI) lower than 25 kg/m².
* Physically active subjects (≥150 min/week of moderate exercise).
* Healthy men and women without neurological, cardiometabolic, immunological, or physical conditions that prevent them from performing physical exercise.
* Participants capable of performing the tests.

Exclusion Criteria:

* History of neuromuscular, cardiac, or diseases that could affect liver or muscle metabolism.
* Use of drugs or other stimulants that interfere with caffeine intake and intestinal absorption during the tests and study.
* Body mass index (BMI) ≥ 25 kg/m².
* Having undergone prolonged periods of forced physical inactivity during the 6 months prior to the study.
* Performing strenuous exercise within 48 hours prior to the tests.
* Failing to replicate the same food intake on the two experimental days.
* Consuming caffeine after 6 PM on the day prior to training or testing.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
cyp1a2 polymorphism | Before the beginning of the trial
  Using saliva sample and PCR
Mean velocity at different %1RM | Through study completion, an average of 2 weeks
  Measuring bar mean velocity desplacement during bench press and back squat exercises.
Peak velocity at different %1RM | Through study completion, an average of 2 weeks
  Measuring bar peak velocity and time to reach peak velocity of bar desplacement during bench press and back squat exercises.
Mean power output at different %1RM | Through study completion, an average of 2 weeks
  Measuring during bench press and back squat exercises.
Peak power output and time to reach peak power output at different %1RM | Through study completion, an average of 2 weeks
  Measuring during bench press and back squat exercises.
Number of repetitions performed in 1 set at 65%1RM until task failure | Through study completion, an average of 2 weeks
  In bench press and back squat exercises
Bar velocity deplacement performed in 1 set at 65%1RM until task failure | Through study completion, an average of 2 weeks
  In bench press and back squat exercises
Power output generated in 1 set at 65%1RM until task failure | Through study completion, an average of 2 weeks
  In bench press and back squat exercise
Maximal Fat Oxidation Rate (MFO) | Through study completion, an average of 2 weeks
  g/min (MFO) using a metabolic chart.
Resting Metabolic Rate (RMR) | Through study completion, an average of 2 weeks
  Kcal at rest (RMR) using a metabolic chart.

SECONDARY OUTCOMES:
Mood state (tension, depression, anger, vigor, fatigue and confusion) | Through study completion, an average of 2 weeks
  Participants graded a set of 29 items related to the mood on a Likert scale from 0 (not at all) to 4 (extremely) in reply to the question: How do you feel at this moment? to assess six scales: tension, depression, anger, vigor, fatigue and confusion.
Adverse effects | Through study completion, an average of 2 weeks
  perception of power, endurance, energy and exertion, as well as heart, muscular and gastrointestinal discomfort
handgrip and isometric mid-thigh pull tests | Through study completion, an average of 2 weeks
  N generated
Vertical Jump (cm) | Through study completion, an average of 2 weeks
Vertical Jump (power) | Through study completion, an average of 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Medicina y Ciencias de la Salud. Universidad de Alcalá, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes